CLINICAL TRIAL: NCT02830906
Title: Comparison of Ramosetron With Ondansetron for Prevention of Intrathecal Morphine Induced Nausea and Vomiting After Primary Total Knee Arthroplasty: A Randomized Control Trial
Brief Title: Effect of Ramosetron in Prevention of Intrathecal Morphine Induced Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, piya pinsornsak, associate professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTC-EC-OT-2-169/56
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Total Knee Arthroplasty; Intrathecal Morphine; Ramosetron; Ondansetron; postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramosetron group (Experimental): Patients received 0.3 mg of intravenous ramosetron before spinal anesthesia and intrathecal morphine
  Interventions: Drug: ramosetron
- ondansetron group (Active Comparator): Patients received 8 mg of intravenous ondansetron before spinal anesthesia and intrathecal morphine
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: ramosetron — intravenous ramosetron 0.3 mg before spinal anesthesia and intrathecal morphine
  Other Names: ramosetorn
  Arms: ramosetron group
Drug: Ondansetron — intravenous ondansetron 8 mg before spinal anesthesia and intrathecal morphine
  Arms: ondansetron group

SUMMARY:
We would like to know the prophylactic anti-emetic effect of ramosetron compare to ondansetron in patient undergone total knee arthroplasty with spinal anesthesia and intrathecal morphine .

DETAILED DESCRIPTION:
The patients were allocated into 2 groups by computerized block randomization according to a computer generated randomization. Treatment allocations were contained in sealed envelopes that were opened after patient enrollment. Patients received either 8 mg of intravenous (IV) ondansetron or 0.3 mg of IV ramosetron 10 minutes before spinal anesthesia and intrathecal morphine. All of the unilateral TKAs were done by one orthopedic surgeon using the same minimally invasive surgical technique and the same prosthesis.

Patients were monitored for incidence of Post Operative Nausea Vomiting(PONV) every 6 hours until 24 hours, and 24-48 hours postoperatively. Common adverse drug reactions associated with serotonin receptor antagonists (pruritus, dizziness, and headache) were also recorded.

The sample size calculation was based on the ability to detect a difference in incidence of postoperative nausea in between the two groups of 40% i.e. 50% in the ondansetron arm, and 30% in the ramosetron arm, consistent with a previous study. Using a power of 80% (β=0.2) and a two sided significance level(alpha) of 0.05, 45 patients in each group were required.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-80 years with a diagnosis of primary OA undergoing unilateral TKA
* American Society of Anesthesiologist (ASA) physical status I-III
* Giving written informed consent

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m2
* Unable to undergo spinal anesthesia
* History of allergic to study drugs
* Impaired renal and/or hepatic function
* Use of systemic steroids and anti-emetics within 24 hours of operation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of postoperative nausea and vomiting | 48 hours after the operation

SECONDARY OUTCOMES:
number of patients require for anti-emetic medicine | 48 hours after the operation
visual analog scale for pain | 48 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: piya pinsornsak, md, Principal Investigator — Thammasat University

IPD SHARING:
Plan to Share IPD: No